CLINICAL TRIAL: NCT01281150
Title: A Phase 1 Study of ABT-888 (Veliparib) in Combination With Weekly Carboplatin and Paclitaxel in Advanced Solid Tumors
Brief Title: Veliparib in Combination With Carboplatin and Paclitaxel in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02490; NCI-2011-02490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000693333; 09-084 (Other: University of Pittsburgh Cancer Institute (UPCI)); 8620 (Other: CTEP); P30CA047904 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Adult Solid Neoplasm; Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; Male Breast Carcinoma; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; veliparib

ARMS (1):
- Treatment (veliparib, paclitaxel, carboplatin) (Experimental): DOSE-ESCALATION: Patients receive veliparib PO twice daily BID on days 1-5, 8-12, and 15-19 and paclitaxel IV over 1 hour and carboplatin IV over 30 minutes in course 1 and 3 hours in subsequent courses on days 3, 10, and 17. After 4 courses, patients receive paclitaxel and carboplatin on days 3 and 10 only. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (Completed as of 12/2012)
  EXPANSION COHORT: Patients receive veliparib PO BID on days 1-21 and paclitaxel IV over 1 hour and carboplatin IV over 3 hours on days 3 and 10. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I clinical trial studies the side effects and the best dose of veliparib when given together with carboplatin and paclitaxel in treating patients with locally advanced or metastatic solid tumors. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by blocking them from dividing. Giving veliparib with carboplatin and paclitaxel may work better in treating patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum-tolerated dose (MTD) of the combination of weekly carboplatin, paclitaxel, and veliparib.

SECONDARY OBJECTIVES:

I. To assess the safety, tolerability, and MTD of the combination of weekly carboplatin, paclitaxel, and veliparib.

II. To assess the safety and toxicity of this combination as determined by the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v. 4.0) and to determine the dose-limiting toxicity (DLT).

III. To determine the pharmacokinetic and pharmacodynamic effects of this combination, including determinations of poly (adenosine diphosphate [ADP]-ribose) polymerase (PAR) in tumor specimens when available, assessment of deoxyribonucleic acid (DNA) damage as measured by gamma H2A histone family, member X (g-H2AX) in skin biopsies and tumor specimens will be obtained.

IV. To assess characteristics of primary tumor specimens that may contribute to efficacy of this combination including breast cancer, early onset (BRCA) by immunohistochemistry, gene analysis of PARP 1, PARP 2, BRCA, and triple negative and homologous recombination repair (HRR) deficiency gene expression signatures.

V. To document any anti-tumor response.

OUTLINE: This is a dose-escalation study of veliparib.

DOSE-ESCALATION: Patients receive veliparib orally (PO) twice daily (BID) on days 1-5, 8-12, and 15-19 and paclitaxel IV over 1 hour and carboplatin IV over 30 minutes in course 1 and 3 hours in subsequent courses on days 3, 10, and 17. After 4 courses, patients receive paclitaxel and carboplatin on days 3 and 10 only. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (Completed as of 12/2012)

EXPANSION COHORT: Patients receive veliparib PO BID on days 1-21 and paclitaxel IV over 1 hour and carboplatin IV over 3 hours on days 3 and 10. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor that has evidence of metastatic spread (stage IV) or is locally advanced and unresectable

  * Patients with breast cancer may have estrogen receptor positive or negative (ER+ or ER-) disease
  * Patients with breast cancer may not be human epidermal growth receptor -2 (HER2)-positive ( 3+), or fluorescent in situ hybridization (FISH) ratio > 2.2
  * Patients in the biopsy expansion cohort must have "triple negative" breast cancer defined as:

    * Estrogen receptor staining < 10%; progesterone receptor staining <10%; Her 2 < 2.2 by FISH, or immunohistochemistry (IHC) 0-2+
* Patients may have been previously treated

  * In the dose escalation cohort, there is no limit to prior therapies
  * In the expansion cohort, patients may have only had 1-3 prior regimens for metastatic disease
  * Patients may have received prior carboplatin, paclitaxel, or poly (ADP-ribose) polymerase (PARP) inhibitor therapy as part of their previous treatment regimens

    * However, patients may NOT have received prior therapy with paclitaxel, carboplatin, and PARP inhibitor in combination
  * Patients must not have received chemotherapy within 4 weeks of starting study (or 6 weeks if prior treatment was with carmustine [BCNU] or mitomycin C)
  * Patients must not have received radiation within 2 weeks of starting study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS)< 2 (Karnofsky > 60%)
* Life expectancy > 2 months
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times ULN
* Creatinine normal within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73m^2 for patients with creatinine levels above institutional normal
* Must able to swallow pills
* Pregnant women are excluded from this study

  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients enrolled in the expanded cohort with mandatory biopsies must:

  * Have accessible tumors
  * Not be on therapeutic anticoagulation
  * Have signed informed consent form

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 2 weeks (4 weeks for central nervous system [CNS] metastases) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib or other agents used in study
* Concurrent treatment with bisphosphonates, or other bone anti-resorptive agent such as denosumab is allowed; concurrent treatment with hormonal therapy (tamoxifen, ovarian suppression with gonadotropin-releasing hormone [GNRH] agonists, aromatase inhibitors) or trastuzumab therapy is NOT allowed in breast cancer patients; prostate cancer patients may continue GNRH agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with veliparib
* Active seizure or history of seizure disorder
* Patients with CNS metastases must be stable after therapy for CNS metastases (such as surgery, radiotherapy or stereotactic radiosurgery) for > 3 months and must be off steroid treatment prior to study enrollment
* Patients who undergo biopsy as part of the study in the expanded dose cohort should not be on anti-coagulants or have a pre-existing coagulopathy
* Peripheral neuropathy of severity greater than grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level one level below the lowest dose where greater than or equal to 2 patients experience a DLT assessed by National Cancer Institute (NCI) CTCAE v. 4.0 | 21 days

SECONDARY OUTCOMES:
Change in BRCA protein levels by immunohistochemistry | Baseline to day 4 of course 2
  Calculated and compared using the Wilcoxon rank sum test.
Change in PAR and g-H2AX in tumor tissue | Baseline to day 4 of course 2
  Assessed with Wilcoxon signed rank tests.
Grade >= 3 non-hematological or any grade 5 DLTs as graded by the NCI CTCAE v. 4.0 | 21 days
  Statistics on the number of cycles received by patients and any dose reductions will be tabulated.
Incidence of adverse events as graded by the NCI CTCAE v. 4.0 | Up to 4 weeks post-treatment
  The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade.
Plasma concentration of carboplatin, paclitaxel, and veliparib using liquid chromatography-mass spectrometry (LC-MS) assay and spectrometry assay | Baseline, at 30 minutes and at 1, 2, 4, and 8 hours on day 3 of course 1
Response complete response [Cr], partial response [PR], and stable disease [SD]) using the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) | Up to 4 weeks post-treatment
  CR, PR, and incidence of SD will be tabulated by disease diagnosis and by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Puhalla, Principal Investigator — University of Pittsburgh Cancer Institute (UPCI)
Locations (3):
- United States (3):
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania